CLINICAL TRIAL: NCT05912790
Title: eyeTube in Combination With the eyeWatch Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rheon Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEN-CL
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Aqueous Humor Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated with the eyeTube (Experimental)
  Interventions: Device: eyeTube

INTERVENTIONS:
Device: eyeTube — Implantation of a drainage device in the eye, in combination with the eyeWatch implant

SUMMARY:
In this study, the investigators want to investigate the success of aqueous humor shunting in the retrobulbar space, using the eyeTube in combination with the eyeWatch implant. The investigators postulate that posterior aqueous humor shunting would be more effective, as this space offers a larger drainage area and a less aggressive local inflammatory environment than the subconjunctival space close to the limbus, resulting in lower and better-sustained IOP than in the more limited, fibroblast-promoting subconjunctival environment surrounding standard implants.

ELIGIBILITY:
Inclusion Criteria:

* - Men and women aged 18 to 85.
* Diagnosis of primary open-angle glaucoma meeting both of the following criteria:
* IOP uncontrolled by at least one (1) or more classes of topical IOP-lowering medical therapy, and
* Failure of at least one (1) conventional intraocular glaucoma surgery (e.g., glaucoma filter surgery or tube shunting) or cilioablative procedures (e.g., cryotherapy, cyclodiode therapy).
* Trabecular meshwork visible on gonioscopy, with a Shaffer angle ≥ 3 in the target quadrant.
* Patients must be able to understand the study requirements and provide written informed consent.
* Patients must be willing to follow study instructions, agree to comply with all study procedures and be able to attend all scheduled follow-up examinations for at least 12 months after surgery.

Exclusion Criteria:

* - Previous filtering surgery, secondary glaucoma, severe systemic disease, pregnancy, breast-feeding, inability to understand or give informed consent.
* Choroidal detachment, choroidal effusion or any active choroidopathy.
* Diagnosis of acute angle-closure glaucoma or malignant glaucoma.
* History of glaucoma drainage/valve implant in target quadrant
* Presence of conjunctival scarring, previous conjunctival surgery or other conjunctival pathology (e.g. pterygium) in the target quadrant.
* Use of systemic (oral or intravenous) glaucoma medications
* History of corneal surgery (including LASIK and PRK), corneal opacities, corneal diseases or any corneal pathology likely to interfere with IOP measurement.
* Eyes with ocular malformations such as microphthalmia
* Eyes with concomitant inflammatory/infectious ocular disorders
* Aphakia
* Presence of an anterior chamber intraocular lens or implantable contact lens
* Previous complicated cataract surgery or presence of vitreous in the anterior chamber
* Cataract surgery performed less than 6 months before the start of the study
* Presence of intraocular silicone oil
* Previous diagnosis of chronic uveitis in either eye
* Active diabetic retinopathy, choroidal neovascularization, secondary retinal vein occlusion, central retinal vein occlusion, proliferative retinopathy or other ophthalmic disease or disorder likely to distort study results.
* Impaired episcleral venous drainage (e.g., Sturge-Weber or nanophthalmos or other evidence of elevated venous pressure)
* Uncontrolled systemic disease (e.g. diabetes, hypertension)
* History of dermatological keloid formation
* Use of ocular or systemic steroids in the last 30 days (chronic continuous use of systemic steroids is permitted) prior to the screening visit, or known response to corticosteroids.
* Pregnant or breast-feeding women, or women of childbearing age who do not wish to use medically acceptable contraception between the screening visit and the 12-month follow-up visit.
* Known or suspected allergy or hypersensitivity to any component of the device (e.g. silicone).
* Current participation or participation within the last 30 days (from the screening visit) in another clinical trial of an investigational drug or interventional device.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) reduction | 12 months
  The proportion of subjects achieving a mean reduction in IOP of ≥ 20% compared with pre-operative pressure at 12 months with the same or fewer hypotensive drugs.
Adverse events | 12 months
  The incidence and severity of adverse events in the study eye (overall and related to the eyeWatch system) throughout the follow-up period.

CONTACTS AND LOCATIONS:
Locations (1):
- Senghor Centre, Mbour, Senegal

IPD SHARING:
Plan to Share IPD: No